CLINICAL TRIAL: NCT02438189
Title: Reduction of Nocturnal Hypoglycemia and Hyperglycemia in the Home Using Predictive Algorithms, Pump Suspension, and Insulin Dosing
Brief Title: Reduction of Nocturnal Hypoglycemia and Hyperglycemia in the Home Using Predictive Algorithms
Acronym: PHM2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PHM2; RFA-DK-08-012 (Other Grant/Funding Number: NIDDK); 5R01DK085591-05 (NIH)
Record Dates: First submitted 2015-05-01; First posted 2015-05-08 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Hypoglycemia; Hyperglycemia; Artificial Pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hyperglycemia Minimization Algorithm (Active Comparator): The hyperglycemia minimization algorithm will be running actively on the study laptop during the night and dose insulin if the algorithm predicts hyperglycemia. If hypoglycemia is predicted, the system will suspend the pump.
  Interventions: Device: Hyperglycemia Minimization Algorithm
- Predictive Low Glucose Suspend (No Intervention): The control algorithm will run passively and not dose additional insulin. If hypoglycemia is predicted, the system will suspend the pump.

INTERVENTIONS:
Device: Hyperglycemia Minimization Algorithm — The hyperglycemia minimization algorithm will be running actively on the study laptop during the night and dose insulin if the algorithm predicts hyperglycemia. If hypoglycemia is predicted, the system will suspend the pump.
  Arms: Hyperglycemia Minimization Algorithm

SUMMARY:
Objective: to gain experience with in-home use of a modified algorithm that will dose insulin to minimize projected hyperglycemia overnight in addition to suspending the pump if hypoglycemia is projected overnight and to obtain feasibility, safety, and initial efficacy data.

Study Design: randomized controlled trial, with randomization on a night level within subject.

Major Eligibility Criteria: clinical diagnosis of type 1 diabetes, daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months; 15.0 to <46.0 years of age; HbA1c < 10.0%; no DKA in last 6 months; no hypoglycemic seizure or loss of consciousness in last 6 months; Living with a significant other or family member ("companion") committed to participating in all study activities, and being present and available to provide assistance when the system is being used at night.

Sample Size: 30 subjects.

Study Duration and Visit Schedule: duration approximately 3 months, with preliminary run-in activities followed by up to 90 days spent in clinical trial phase of study; clinic visits at enrollment, following CGM and system assessment run-in phases, at start of clinical trial phase, at 21-day point of clinical trial phase, and after 42 nights of successful system use.

Major Efficacy Outcomes:

* Primary: time in range (70-180 mg/dl, 3.9-10.0 mmol/L) overnight.
* Secondary: time spent in hypoglycemia (≤70 mg/dl, 3.9 mmol/L) and time spent in hyperglycemia (>180 mg/dl, 10.0 mmol/L) overnight.

Major Safety Outcomes: CGM measures of hypo- and hyperglycemia, including morning blood glucose and mean overnight sensor glucose; adverse events including severe hypoglycemia and diabetic ketoacidosis.

DETAILED DESCRIPTION:
Subjects who are eligible for the clinical trial initially will use a Veo insulin pump and Enlite 2 CGM sensor at home for a minimum of 6 days/week over a 2-week period to verify that the subject is able to use the CGM and insert sensors.

The first 10 subjects enrolled will participate in a 2-day overnight hotel-based pilot, collecting a total of 20 nights of data and experience with the system in a transitional hotel setting. The DSMB will review safety data from the 20 night hotel-based pilot study and make recommendations regarding proceeding to the at-home portion of the study.

Following DSMB review and approval of the safety data from the hotel study, the first 10 subjects will participate in an Algorithm Assessment Phase of approximately 10 nights of Predictive Low Glucose Suspend (PLGS) + Hyper Minimization system use each (for a nominal total of 100 nights of use at home) to determine if any adjustments to the algorithm parameters are needed and if it is safe to advance to the randomized clinical trial phase. If adjustments are needed, the Algorithm Assessment Phase will be repeated, using the same 10 subjects if possible. Once the randomized clinical trial phase begins, approximately 200 nights of randomized system use will be collected and assessed for safety by the DSMB before proceeding.

New subjects who enroll in the study after the completion of the Algorithm Assessment Phase will use the PLGS+Hyper Minimization closed-loop system at home for at least 5 days to demonstrate their ability to use the system and submit study data to the Coordinating Center.

Subjects who successfully demonstrate their ability to use the system at home as described above will be eligible for the randomized trial phase. This phase consists of use of the full system in the home for approximately 42 nights:

* Each night the blood glucose level will be checked with the BG meter and used to perform a calibration of the CGM. This calibration must occur no more than 90 minutes prior to activation of the system. NOTE: Subjects will be instructed to calibrate the CGM per manufacturer guidelines.
* Then the system will be activated, linking the CGM and insulin pump to the computer at the bedside.
* A randomization schedule on the laptop will be used to determine whether the system will run in PLGS+Hyper Minimization mode or PLGS-only.
* Subjects will be blinded as to whether the system is running in PLGS+Hyper Minimization mode or PLGS-only.
* There will not be an alarm if the pump shuts off or if automated insulin dosing occurs. The CGM alarm will be set to 60 mg/dL (3.3 mmol/L). When a CGM alarm occurs, the subject will be asked to measure the blood glucose with a BG meter, if he/she is aware of the alarm.
* The time period for outcome assessment each night will be from the time the system is activated until it is turned off in the morning.
* Pump shut off, when it occurs, will be for up to 120 minutes in a 150-minute period, and no more than 180 minutes for the entire night. Multiple instances of pump suspension can occur if there are recurrent predictions of hypoglycemia during the night.
* Small correction boluses of insulin will be delivered when the system predicts that hyperglycemia above a pre-set threshold will occur, with insulin-on-board constraints and cumulative delivery limits to minimize the likelihood of excessive insulin delivery.
* Subjects will be asked to check blood glucose with the study BG meter each morning prior to breakfast and enter the results using the controller software interface. The subject will be instructed to contact the study physician if the morning blood glucose value is <60 mg/dl (3.3 mmol/L) or >300 mg/dl (16.7 mmol/L). Monitoring processes detailed in section 3.11 will ensure that the subject can be contacted if these values are not reported as required or are out of range.
* Subjects will be asked to record all overnight carbohydrate intake using the controller software interface.
* Subjects will be asked to perform periodic CGM data uploads using the controller software interface. Monitoring processes will ensure that the subject can be contacted if these uploads do not occur as required, or if review of an upload reveals any extreme, prolonged episodes of hypoglycemia or hyperglycemia, or elevated morning blood glucose values.

Upon completion of the study, subjects as well as study clinicians will be asked to complete a human factors usability questionnaire regarding use of the study system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes and using daily insulin therapy for at least one year and an insulin infusion pump for at least 6 months The diagnosis of type 1 diabetes is based on the investigator's judgment; C peptide level and antibody determinations are not required.
* Age 15.0 to <46.0 years
* HbA1c <10.0%

  * Measured with DCA2000 or equivalent device for assessing eligibility
  * HbA1c measurements performed as part of usual clinical care within 2 weeks prior to obtaining informed consent for participation in the trial may be used.
* Uninterrupted internet access while study system is being used overnight and for upload of study data in the morning
* Living with a significant other or family member ("companion") committed to participating in all study activities, and being present and available to provide assistance when the system is being used at night
* An understanding of and willingness to follow the protocol and sign the informed consent

Exclusion Criteria:

* Diabetic ketoacidosis in the past 3 months
* Hypoglycemic seizure or loss of consciousness in the past 6 months
* History of seizure disorder (except for hypoglycemic seizure)
* History of any heart disease including coronary artery disease, heart failure, or arrhythmias
* Cystic fibrosis
* Current use of oral/inhaled glucocorticoids, beta-blockers or other medications, which in the judgment of the investigator would be a contraindication to participation in the study.
* History of ongoing renal disease (other than microalbuminuria). Creatinine level must have been obtained within the last year if subject has diabetes of >10 years duration. If creatinine is >1.5 mg/dL (132 µmol/L), the subject is excluded.
* Medical or psychiatric condition that in the judgment of the investigator might interfere with the completion of the protocol such as:

  * Inpatient psychiatric treatment in the past 6 months
  * Uncontrolled adrenal disorder
  * Abuse of alcohol
* Pregnancy Negative urine pregnancy test required for females who have experienced menarche as well as agreement from subject and parent/guardian to use a form of contraception to prevent pregnancy while participant is in the study. Subjects who become pregnant will be discontinued from the study.
* Liver disease as defined by an ALT greater than 3 times the upper limit of normal

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Comparison of percent time in range overnight between the two treatment arms | Up to 42 nights
  A single percentage calculated for each subject by pooling all CGM readings from the hyperglycemia minimization active algorithm nights will be compared with the corresponding percentage obtained by pooling all of the data from control nights for the same subject. All CGM readings will be weighted equally in the pooled percentage regardless of how they distribute across nights.

SECONDARY OUTCOMES:
Mean CGM glucose overnight | Up to 42 nights
Percentage of time spent with CGM <50 mg/dL (2.8 mmol/L) | Up to 42 nights
Percentage of time spent with CGM <60 mg/dL (3.3 mmol/L) | Up to 42 nights
Percentage of time spent with CGM <70 mg/dL (3.9 mmol/L) | Up to 42 nights
Percentage of time spent with CGM >180 mg/dL (10.0 mmol/L) | Up to 42 nights
Percentage of time spent with CGM >250 mg/dL (13.9 mmol/L) | 42 nights
Percentage of time spent with CGM >300 mg/dL (16.7 mmol/L) | Up to 42 nights
Percentage of nights with >30 min and >60 min consecutive CGM values <50 mg/dL (2.8 mmol/L) | Up to 42 nights
Percentage of nights with >30 min and >60 min consecutive CGM values <60 mg/dL (3.3 mmol/L) | Up to 42 nights
Percentage of nights with >30 min and >60 min consecutive CGM values <70 mg/dL (3.9 mmol/L) | Up to 42 nights
Glucose coefficient of variation (CV) | Up to 42 nights
Amount of total insulin boluses | Up to 42 nights
Mean home glucose meter morning glucose | Up to 42 nights
Morning glucose measured with home glucose meter >250 mg/dL (13.9 mmol/L) | Up to 42 nights
Mean sensor glucose over 24 hours | Up to 42 nights
Mean sensor glucose 4 hours post system deactivation | Up to 42 nights
Percentage of sensor glucose values 70 to 180 mg/dL (3.9 to 10.0 mmol/L) overnight | Up to 42 nights
Percentage of sensor glucose values 70 to 180 mg/dL (3.9 to 10.0 mmol/L) 4 hours after system deactivation | Up to 42 nights
Percentage of sensor glucose values 70 to 180 mg/dL (3.9 to 10.0 mmol/L) over 24 hours | Up to 42 nights
Change in HbA1c from clinical baseline to study completion | Up to 42 nights

CONTACTS AND LOCATIONS:
Overall Officials: Roy Beck, MD, PhD, Principal Investigator — Jaeb Center for Health Research; Bruce Buckingham, MD, Study Chair — Stanford University; John Lum, MS, Study Director — Jaeb Center for Health Research
Locations (3):
- United States (2):
  - Stanford University, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Spaic T, Driscoll M, Raghinaru D, Buckingham BA, Wilson DM, Clinton P, Chase HP, Maahs DM, Forlenza GP, Jost E, Hramiak I, Paul T, Bequette BW, Cameron F, Beck RW, Kollman C, Lum JW, Ly TT; In-Home Closed-Loop (IHCL) Study Group. Predictive Hyperglycemia and Hypoglycemia Minimization: In-Home Evaluation of Safety, Feasibility, and Efficacy in Overnight Glucose Control in Type 1 Diabetes. Diabetes Care. 2017 Mar;40(3):359-366. doi: 10.2337/dc16-1794. Epub 2017 Jan 18. PMID 28100606